CLINICAL TRIAL: NCT02878564
Title: Effect of Schistosomiasis Mansoni and Its Treatment on HIV Susceptibility and Female Genital Immunology
Brief Title: Effect of Schistosomiasis Mansoni on HIV Susceptibility and Female Genital Immunology
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: UVRI-IAVI HIV Vaccine Program, Uganda (Unknown)
Responsible Party: Principal Investigator, Rupert Kaul, Professor, University of Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UT-Schisto
Record Dates: First submitted 2016-08-15; First posted 2016-08-25 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Schistosomiasis Mansoni; HIV
Keywords: Schistosomiasis mansoni; HIV susceptibility; Genital immunology; Mucosal immunology; HIV entry assay; Adult women
MeSH Terms: conditions — Schistosomiasis mansoni | interventions — Praziquantel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Praziquantel treatment (Experimental): Participants will be HIV-uninfected women with asymptomatic Schistosoma mansoni infection; the study will examine the impact of standard praziquantel therapy (40 mg/kg po single dose) on genital immunology and HIV susceptibility.
  Interventions: Drug: Praziquantel

INTERVENTIONS:
Drug: Praziquantel — 40 mg/kg, PO (orally administered tablets)
  Other Names: Agopraz, bromoxel, biltricide

SUMMARY:
The aim of this study is to assess the impact of Schistosoma mansoni infection and its treatment on genital immunology and HIV susceptibility in Ugandan women.

DETAILED DESCRIPTION:
Schistosomiasis mansoni is a water-borne disease caused by helminth Schistosoma mansoni (S. mansoni), in which adult worms deposit eggs in mesenteric blood vessels. Schistomiasis prevalence in the fishing communities in East Africa, and particularly in the Lake Victoria region, exceeds 60% and there is overlap in this region with a high prevalence of HIV (29%).

A recent epidemiological study found an association between S. mansoni and HIV infection in adult women residing near Lake Victoria in Tanzania. Furthermore, in primate studies S. mansoni infection was shown to increase susceptibility to SIV infection after rectal (but not intravenous) challenge, implying that S. mansoni might increase HIV susceptibility by altering local mucosal (gut) immunology.

While S. mansoni does not directly infect the genital tract, we hypothesize that the inflammation it causes in the gut may be associated with mucosal inflammation at other sites through activation of common mucosal homing integrins such as a4b7. Therefore in this study we propose to explore whether S. mansoni increases inflammation and/or HIV susceptibility in the endocervix of adult women.

HIV-uninfected adult women from Entebbe, Uganda will be screened for schistosomiasis using a commercial CCA rapid test kit, and infected women who fulfill the study eligibility criteria will be recruited into the study. Kato-Katz microscopy analysis will be performed to assess egg shedding at baseline. Additionally, urine microscopy will be done to screen for Schistosoma hematobium (which can directly involve the genital mucosa). Schistosomiasis treatment will be provided to all participants according to Ugandan clinical guidelines.

Endocervical cytobrush, vaginal SoftCup and blood samples will be collected at three time points; at baseline and 4 and 8 weeks after schistosomiasis treatment, at the same stage of the menstrual cycle. Using an ex vivo HIV entry assay and mucosal cytokine and microbiome analyses we will quantify the effect of S. mansoni and its treatment on cervical HIV susceptibility and genital inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Positive (score above "trace") on a urine CCA rapid test
* Willing to be treated with praziquantel
* Willing to give informed consent, and answer short questionnaires on economic status, and sexual risk behavior.
* Willing to comply with the requirements of the protocol
* HIV and classical STI (see below) negative

Exclusion Criteria:

* HIV infected
* Malaria infected
* Pregnant.
* Irregular menstrual cycle, or actively menstruating at the time of genital sampling.
* Tested positive for classical STIs (syphilis, gonorrhea, chlamydia, Trichomonas vaginalis) or having genital ulcers
* Prior hysterectomy
* Deemed by physician to be unlikely to complete study protocol.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2016-03; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change in the percentage of endocervical CD4+ T cells susceptible to HIV pseudovirus entry after treatment of schistosomiasis. | 1 month.
  The percentage of endocervical CD4+ T cells per cytobrush infected ex vivo by an HIV pseudovirus construct, as quantified by flow cytometry.
Change in the number of endocervical CD4+ T cells susceptible to HIV pseudovirus entry after treatment of schistosomiasis. | 1 month.
  The number of endocervical CD4+ T cells per cytobrush infected ex vivo by an HIV pseudovirus construct, as quantified by flow cytometry.

SECONDARY OUTCOMES:
Change in the percentage of blood CD4+ T cells susceptible to HIV pseudovirus entry after treatment of schistosomiasis. | 1 and 2 months.
  The percentage of blood CD4+ T cells infected ex vivo by an HIV pseudovirus construct, as quantified by flow cytometry.
Change in the phenotype of endocervical and blood CD4+ T cells after treatment of schistosomiasis. | 1 and 2 months.
  Surface expression of CCR5, CD69, CD38, HLA-DR, a4b7, CCR7 and CD45RA by endocervical and blood CD4 T will be assessed using flow cytometry.
Change in genital proinflammatory cytokine levels after treatment of schistosomiasis. | 1 and 2 months.
  A predefined genital inflammation score based on genital levels of pro-inflammatory cytokines and chemokines [as per Arnold K et al, Muc Immunol, 2015] will be assessed.
Change in the cervico-vaginal microbiome after treatment of schistosomiasis. | 1 and 2 months.
  The cervico-vaginal microbiome will be assessed by 16s rRNA sequencing before and after schistosomiasis therapy.
Change in the cervico-vaginal proteome after treatment of schistosomiasis. | 1 and 2 months.
  The genital proteome will be assessed by mass spectrometry before and after schistosomiasis therapy.
Change in the percentage of endocervical CD4+ T cells susceptible to HIV pseudovirus entry after treatment of schistosomiasis. | 2 months.
  The percentage of endocervical CD4+ T cells per cytobrush infected ex vivo by an HIV pseudovirus construct, as quantified by flow cytometry.
Change in the number of endocervical CD4+ T cells susceptible to HIV pseudovirus entry after treatment of schistosomiasis. | 2 months.
  The number of endocervical CD4+ T cells per cytobrush infected ex vivo by an HIV pseudovirus construct, as quantified by flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Rupert Kaul, MD/PhD, Principal Investigator — University of Toronto
Locations (1):
- UVRI-IAVI HIV Vaccine program, Entebbe, Wakiso, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arnold KB, Burgener A, Birse K, Romas L, Dunphy LJ, Shahabi K, Abou M, Westmacott GR, McCorrister S, Kwatampora J, Nyanga B, Kimani J, Masson L, Liebenberg LJ, Abdool Karim SS, Passmore JA, Lauffenburger DA, Kaul R, McKinnon LR. Increased levels of inflammatory cytokines in the female reproductive tract are associated with altered expression of proteases, mucosal barrier proteins, and an influx of HIV-susceptible target cells. Mucosal Immunol. 2016 Jan;9(1):194-205. doi: 10.1038/mi.2015.51. Epub 2015 Jun 24. PMID 26104913
- [Background] Downs JA, van Dam GJ, Changalucha JM, Corstjens PL, Peck RN, de Dood CJ, Bang H, Andreasen A, Kalluvya SE, van Lieshout L, Johnson WD Jr, Fitzgerald DW. Association of Schistosomiasis and HIV infection in Tanzania. Am J Trop Med Hyg. 2012 Nov;87(5):868-73. doi: 10.4269/ajtmh.2012.12-0395. Epub 2012 Oct 1. PMID 23033399
- [Background] Chenine AL, Shai-Kobiler E, Steele LN, Ong H, Augostini P, Song R, Lee SJ, Autissier P, Ruprecht RM, Secor WE. Acute Schistosoma mansoni infection increases susceptibility to systemic SHIV clade C infection in rhesus macaques after mucosal virus exposure. PLoS Negl Trop Dis. 2008 Jul 23;2(7):e265. doi: 10.1371/journal.pntd.0000265. PMID 18648516
- [Background] Joag VR, McKinnon LR, Liu J, Kidane ST, Yudin MH, Nyanga B, Kimwaki S, Besel KE, Obila JO, Huibner S, Oyugi JO, Arthos J, Anzala O, Kimani J, Ostrowski MA; Toronto HIV Research Group; Kaul R. Identification of preferential CD4+ T-cell targets for HIV infection in the cervix. Mucosal Immunol. 2016 Jan;9(1):1-12. doi: 10.1038/mi.2015.28. Epub 2015 Apr 15. PMID 25872482